CLINICAL TRIAL: NCT01743170
Title: Leuven Academic Programme for Telemonitoring of Hypertensive Patients
Brief Title: Telemonitoring of Hypertensive Patients
Acronym: LAPTOHP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment by GPs proved to be impossible
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Jan A. Staessen, Professor of Medicine, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAPTOHP
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: Blood pressure control; Hypertension; Office blood pressure; Self-measured blood pressure; Telemonitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): In the control group doctors will receive information on the self-measured blood pressure as recorded at home via a diary card.
- Intervention group (Experimental): In the intervention group, doctors will receive weekly reports via telemonitoring of self-measured blood pressure.
  Interventions: Other: Telemonitoring of self-measured blood pressure

INTERVENTIONS:
Other: Telemonitoring of self-measured blood pressure — In the intervention group, doctors receive weekly reports via telemonitoring on the self-measured blood pressure
  Arms: Intervention group

SUMMARY:
The proportion of hypertensive patients achieving adequate blood pressure control meeting guideline targets remains low. Of hypertensive patients, only 50% are on antihypertensive medications. Of those on blood pressure lowering drugs, only 50% have their blood pressure controlled.

The objectives of this study are:

1. To test the feasibility of telemonitoring of blood pressure in Flemish general practices.
2. To investigate in a randomized fashion whether telemonitoring enabled self-measurement of blood pressure leads to faster blood pressure control than self-measurement without the telemonitoring information.
3. The secondary endpoints include various blood pressure indexes, adverse effects, a simple assessment of quality of life, adherence, a log of technical problems, and cost effectiveness (EQ-5D-5L).

DETAILED DESCRIPTION:
Hypertension affects an estimated 20% to 30% of the world's adult population. Despite the availability of numerous safe and effective pharmacologic therapies, including single-pill combinations of 2-3 drugs, the percentage of patients achieving adequate blood pressure control meeting guideline targets remains low. The rule of halves still applies. Of hypertensive patients, only 50% are on antihypertensive medications. Of those on blood pressure lowering drugs, only 50% have their blood pressure controlled. Achieving target blood pressure levels in the treatment of hypertension requires that patients take their medications not only properly (adherence), but also continue to do so throughout long-term treatment (persistence). Poor medication-taking behavior is a major problem among patients with hypertension, and is one of the main causes of failure to achieve blood pressure control. Self-measurement of blood pressure at home improves adherence to treatment and the control of blood pressure. One might even hypothesize that telemonitoring of blood pressure, which allows instantaneous feedback between doctor and patient might even be more effective than usual self-measurement in improving adherence and reaching treatment tools.

Previous studies demonstrated the feasibility of telemonitoring of blood pressure. However, several issues remain unaddressed.

* Feasibility of telemonitoring within the Belgian context has never been tested. No attempt has ever been made in Belgium to assess adherence to antihypertensive drugs in primary care.
* Telemonitoring of blood pressure will never make it to the routine clinical practice unless it can be proven that application of the technique results in faster and better blood pressure control compared with usual care including self-measurement of blood pressure at home.
* Secondary endpoints must also include adverse events, a simple assessment of quality of life, adherence, a log of technical problems, and cost-effectiveness.

LAPTOHP is a randomized parallel-group study, which will address the feasibility and potential benefits of telemonitoring of blood pressure at home. Eligible patients will be recruited at seven general practices. LAPTOHP will include three stages

* Screening period followed by stratification and randomization: Screening involves checking inclusion and exclusion criteria, ruling out secondary hypertension remediable by specific treatment, and obtaining informed written consent as outlined in the Helsinki declaration. Eligible patients will be stratified by centre and randomized in a one-to-three proportion to control or intervention. Randomization will be implemented by sequentially numbered sealed envelopes, which contain the group assignment. These envelopes will be available at the practices, so that no contact with the Studies Coordinating Centre (SCC) will be necessary to randomize the patient.
* Randomised period: Investigators will optimize medical treatment by rotating patients through different classes of antihypertensive drugs, combining drug classes according to the current guidelines of the European Societies of Cardiology and Hypertension (ESC/ESH), while achieving the maximal tolerated dose of each drug. In the intervention group, investigators will receive a report on the telemonitoring data at weekly intervals; in the control group doctors will receive information on the self-measured blood pressure as recorded at home in the week preceding the office visit via a diary card. Doctors are free to schedule contacts with their patients and office visits at their own discretion or as indicated by the clinical context. Once blood pressure control is achieved, the blood pressure measuring devices (telemonitoring enabled or not) will be recuperated and will become available for a next patient. In the control group, patients will keep a diary card in the week preceding the office visits. In the control group, doctors will receive a full report on all telemonitoring data at the completion of randomized treatment, after patients have achieved blood pressure control.
* Late follow-up: Three months after achieving blood pressure control, all patients will be telemonitored for 1 week and complete a diary card, preceding an office visit.

ELIGIBILITY:
Inclusion Criteria:

* Women and men are eligible. Women of reproductive age should apply effective contraception.
* Age ranges from 20 years (inclusive) to less than 80 years.
* Patients should have hypertension, which is uncontrolled on medical treatment.
* At the screening visit, patients should either be untreated for at least 4 weeks or taking a stable drug regimen for at least 4 weeks.
* Medical treatment can consist of all major drug classes. This includes diuretics, β-blockers, α-blockers, calcium-channel blockers (CCBs), inhibitors of the rennin system (angiotensin-converting enzyme inhibitors (ACEIs), angiotensin II type-1 receptor blockers (ARBs), the direct renin inhibitor aliskiren, aldosterone receptor antagonists (ARAs) centrally acting antihypertensive drugs and vasodilators (hydralazine). In line with current recommendations and recent studies, unless contra-indicated or not tolerated, aldosterone antagonists, such as spironolactone 25 to 50 mg per day should have been attempted for at least 4 weeks to improve blood pressure control in treatment-resistant patients.
* The patients should be intellectually and emotionally capable of measuring their blood pressure at home and accept to keep a diary (control group) or to have a report sent to their doctor (intervention group).
* Patient should provide written informed consent.

Exclusion Criteria:

* The clinical context is suboptimal for telemonitoring of blood pressure:

  * Myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 6 months of the screening period.
  * Type-1 diabetes mellitus requiring multiple adjustments of treatment to maintain control or diabetes mellitus with recent hyperglycemic or hypoglycemic coma.
  * Renal dysfunction defined as an estimated glomerular filtration rate (eGFR) of less than 30 mL/min/1.73m², using the Modification of Diet in Renal Disease (MDRD) formula.
  * Secondary hypertension, in which treatment options other than antihypertensive drug treatment are indicated.
  * Sleep apnea syndrome that qualifies for treatment with continuous positive airway pressure (CPAP).
  * Atrial fibrillation or arrhythmia making oscillometric blood pressure measurement unreliable.
  * The patient is on a waiting list for elective surgery or a cardiovascular intervention.
  * Patients with alcohol or substance abuse or psychiatric illnesses.
* The patients should not have any serious medical condition, which in the opinion of the investigator, may adversely interfere with self-measurement of blood pressure at home.
* Patients should not participate in any other trial of an investigational drug or device.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to blood pressure control | During the treatment period, there will be no fixed interval between visits, so that doctors can apply their routine care scheme. Expected average of 3 months.
  Blood pressure control will be defined as a self-measured blood pressure at home below 135 mm Hg systolic and 85 mm Hg diastolic. Blood pressure control is assumed to be present if the aforementioned levels are attained during the week preceding the last office visit of the randomized treatment visit.

SECONDARY OUTCOMES:
Proportion of patients reaching blood pressure control on self-measurement at home and office measurement. | During treatment period. No fixed time interval between visits. Expected average of 3 months.
  Blood pressure control on office measurement is a seated blood pressure below 140 mm Hg systolic and 90 mm Hg.
The proportion of patients reaching and maintaining blood pressure control on self-measurement and office measurement at the late follow-up visit. | Three months after achieving blood pressure control
  A self-measured home blood pressure of less than 135 mmHg systolic and less than 85 mmHg diastolic
The intensity of medical treatment. | During treatment period, up to 3 months.
  The number of antihypertensive drug classes
Adverse events | During treatment period, up to 3 months.
  Adverse events will be recorded by a self-administered questionnaire (as in previous studies conducted in general practice in Belgium).
Assessment of drug adherence. | During treatment period, up to 3 months.
  The Morisky questionnaire will be used to assess drug adherence.
Assessment of quality of life | During treatment period, up to 3 months.
  The EQ-D5 questionnaire will be used for the assessment of quality of life.
Analysis of cost-effectiveness | After completion of the study (expected average is 3 months).
  The cost-effectiveness analysis will be conducted from the perspective of the Belgian health care system, including both the direct and indirect costs of the intervention. The costs will be balanced against the use of medical resources, including visits, medications, and use of medical resources.

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Staessen, MD, PhD, Principal Investigator — University of Leuven
Locations (7):
- Belgium (7):
  - Center C2, Boutersem
  - Center C3, Grimde
  - Center C4, Leuven
  - Center C6, Leuven
  - Center C7, Leuven
  - Center C5, Tienen
  - Center C1, Wilsele